CLINICAL TRIAL: NCT06649487
Title: Investigation of the Effect of Hypertension on Hemodynamics in the Prone Position
Brief Title: Effect of Hypertension on Hemodynamics in the Prone Position
Status: Enrolling by invitation | Type: Observational
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Ali Genc, Assistant professor, Tokat Gaziosmanpasa University
Other Study IDs: 24-KAEK-216
Record Dates: First submitted 2024-10-16; First posted 2024-10-18 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Hypertension; Disk Herniation
Keywords: Anesthesia, General; Prone Position; Hemodynamic Monitoring
MeSH Terms: conditions — Hypertension; Intervertebral Disc Displacement

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Long-term use of antihypertensive drugs in patients diagnosed with hypertension may cause sharp fluctuations in the patient's hemodynamic values such as blood pressure during anesthesia. Low blood pressure that occurs during surgery may cause serious organ failure and even death, especially in patients in the prone position.

These conditions resulting from hypotension increase with prolonged exposure to hypotension. Therefore, it is very important to predict and prevent hypotension in spinal surgery.

In patients with hypertension, the prone position may cause some hemodynamic changes compared to those without comorbidities. Therefore, in this study, researchers planned to investigate the changes in some hemodynamic values in patients with hypertension and without comorbidities who were scheduled for spinal surgery.

DETAILED DESCRIPTION:
The number of spine surgeries has increased in recent years due to degenerative diseases of the spine and age. Lumbar spine surgery is a surgery performed in the prone position. Changing the patient's position from supine to prone may cause a decrease in cardiac output, arterial pressure and tissue perfusion due to the decrease in the preload of the heart. In addition to the decrease in venous return due to increased intra-abdominal pressure, left ventricular compliance may be impaired due to increased thoracic pressure. All these changes may cause decreased cardiac output and systemic hypotension. These changes may be more pronounced especially with the prone position accompanied by anesthesia. This situation is thought to be due to the fact that anesthetic drugs cause direct hypotension as well as impairing reflex responses to hypotension such as the sympathetic system. Perioperative cardiac complications are the main causes of mortality after non-cardiac surgery. Intraoperative hypotension, especially in patients in the prone position, has been shown to be significantly associated with clinical outcomes such as spinal cord ischemia and postoperative vision loss and may lead to serious complications. Therefore, optimization of hemodynamic variables is an integral part of perioperative care to reduce postoperative mortality and morbidity during surgeries that require patients to be placed in the prone position, such as vertebral surgery.

More than 280 million surgeries are performed worldwide each year, and approximately one-third of these patients use antihypertensive agents before surgery. It has been reported that hypertension is associated with hypotension, especially after induction, in patients receiving general anesthesia. Therefore, it has been stated that perioperative management of patients receiving antihypertensive drugs is especially important. Patients diagnosed with preoperative hypertension have been associated with increased risk of surgical bleeding, stroke, and cardiovascular complications. Long-term use of antihypertensive drugs in hypertensive patients may cause autonomic nerve dysfunction, leading to perioperative hypovolemia, decreased tolerance to postural changes, and sharp fluctuations in circulation. Therefore, maintaining hemodynamic stability in hypertensive patients receiving general anesthesia may be difficult. The change in prone position required for vertebral surgery may be associated with a high risk of developing hypotension due to decreased venous return from inferior vena cava compression and increased intrathoracic pressure. In awake patients, hypotension caused by changes in position is prevented by baroreceptor reflex and sympathetic activation, whereas in anesthetized patients, anesthetic drugs may block these compensatory mechanisms, potentially increasing the incidence of hypotension associated with postural change. It has been reported that the incidence of hypotension associated with the change from supine to prone position under general anesthesia is approximately three times higher than in awake patients. However, there are also studies reporting that perioperative hemodynamic changes in patients with hypertension are similar to those without additional comorbidities. MostCare (Vytech Health™, Vygon, Padova, Italy) is a self-calibrating device based on continuous analysis of the systolic and diastolic phases of the arterial waveform via an intraarterial catheter. In short, this monitoring method provides valuable information in terms of cardiac and vascular functions and intravascular volume, as well as close monitoring of blood pressure. It is an important guide in the rapid recognition of etiology and treatment of hemodynamic changes. Spine surgery is mostly performed in the prone position and under general anesthesia. Both general anesthesia and prone position can cause significant changes in the patient's hemodynamics. However, there are limited studies on hemodynamic changes during anesthesia of patients diagnosed with hypertension, and their results are contradictory. In this study, researchers aimed to investigate the effect of hypertension on cardiovascular and hemodynamic changes in the prone position.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ASA scores between 1 and 3 who wish to participate in the study.
* Patients between the ages of 18-75 who are scheduled for vertebral surgery

Exclusion Criteria:

* Heart failure
* Severe arrhythmia
* Severe respiratory failure
* Renal failure
* Chronic liver disease
* Moderate and severe anemia
* Severe fluid and electrolyte disturbances
* Uncontrolled hypertension (systolic blood pressure ≥ 180 mmHg or diastolic blood pressure ≥ 100 mmHg)
* Severe thyroid dysfunction
* Advanced psychiatric illness.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Prone position may cause some hemodynamic changes in patients with hypertension compared to those without comorbidities. Therefore, in this study, researchers planned to investigate the changes in some hemodynamic values in patients with hypertension and without comorbidities who were scheduled for vertebral surgery.
  When calculating the sample size; a previous study has shown that the cardiac index is 2.5±0.3 with a change in prone position under general anesthesia. By estimating a change of approximately 10% in this value in patients with hypertension, when the type 1 error value is accepted as 0.05 and the power is 0.90, it has been determined that the sample size for the study is sufficient with 64 patients. Considering the losses that may occur during follow-up, it is planned to conduct the study with 70 patients with a 10% increase.
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Cardiac output | Hemodynamic parameters will be recorded 1 minute before prone position (T1), 1 minute after prone position (T2), 5 minutes after prone position (T3), 15 minutes after prone position (T4), 30 minutes after prone position (T5) and skin incision time (T6).
  Cardiac output is how many liters of blood heart pumps in one minute.

SECONDARY OUTCOMES:
Blood pressure (systolic, diastolic and mean) | Hemodynamic parameters will be recorded 1 minute before prone position (T1), 1 minute after prone position (T2), 5 minutes after prone position (T3), 15 minutes after prone position (T4), 30 minutes after prone position (T5) and skin incision time (T6).
  Systolic pressure is the maximum blood pressure during contraction of the ventricles; diastolic pressure is the minimum pressure recorded just prior to the next contraction. The mean arterial pressure (MAP) is the average arterial pressure throughout one cardiac cycle, systole, and diastole. The unit of measurement of blood pressure is mmHg.

CONTACTS AND LOCATIONS:
Locations (1):
- Tokat Gaziosmanpasa University, Tokat Province, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided